CLINICAL TRIAL: NCT02802540
Title: Nabilone Effect on the Attenuation of Anorexia, Nutritional Status and Quality of Life in Patients With Anorexia Associated With Advanced Lung Cancer: Randomized Double Blind Clinical Trial
Brief Title: Nabilone Effect on the Attenuation of Anorexia, Nutritional Status and Quality of Life in Lung Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez MD, MD M Sc, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NABILONA
Record Dates: First submitted 2016-05-22; First posted 2016-06-16 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Non-Small Cell Lung Cancer; Anorexia; Cachexia; Weight Lose
Keywords: nabilone; anorexia; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Anorexia; Cachexia | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nabilone (Experimental): Patients start receiving a dose of 0.5 mg daily oral nabilone the first 2 weeks and then 1 mg to complete 8 weeks.
  Interventions: Drug: Nabilone
- placebo (Placebo Comparator): Patients start receiving a dose of 0.5 mg daily oral placebo the first 2 weeks and then 1 mg to complete 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabilone — Patients going to take 0.5 mg capsules of nabilone (CESAMET) the first 2 weeks and then increased to 1 mg to complete 8 weeks.
  Other Names: cesamet
  Arms: Nabilone
Drug: Placebo — Patients going to take capsules of placebo until complete 8 weeks.
  Other Names: placebo nabilona
  Arms: placebo

SUMMARY:
Anorexia is common symptom in cancer patients and is associated with increased morbidity and mortality. However timely detection with objective tools is necessary to establish the diagnosis of anorexia and to assess the magnitude of change over time. The anorexia pathophysiology is not clearly understood and treatment options are limited. Anecdotal historical benefits of smoking marijuana on nausea, pain and anorexia led to studies with marijuana and synthetic cannabinoids from Δ-9-tetrahydrocannabinol, the main active agent in marijuana. The endogenous cannabinoid system with its receptors CB1 and CB2 regulate appetite in four functional levels: (1) limbic system (hedonistic quality), (2) hypothalamus (appetite stimulant), (3) intestinal, and (4) tissue adipose.

Nabilone, a synthetic analogue of THC approved in Mexico for nausea and vomiting induced by chemotherapy is also used in palliative care units for clinical improvement in increased appetite patients in terminal stages, however, there are no clinical trials demonstrating this benefit.

DETAILED DESCRIPTION:
Background: Lung cancer is the leading cause of cancer death in Mexico and the world. Malnutrition is often associated with this type of cancer appearing in about 40-50% of patients the diagnosis made, affecting the quality of life and prognosis, as well as increased toxicity to cancer treatment. Cancer anorexia is characterized by loss of appetite and is the main cause of reduced food consumption in lung cancer patients. Anorexia occurs in up to 25% of cases. Unfortunately, current therapies available to treat anorexia and / or cachexia associated with cancer provide only partial results, mainly because the intervention is delayed and the development of an early and effective intervention is still looking.

In most patients, malnutrition is associated with a hyporexia secondary to the production of pro-inflammatory cytokines such as tumor necrosis factor (TNF), leading to an increase in metabolism and appetite loss. Nabilone is a synthetic cannabinoid derivative that is widely used in oncology for its antiemetic and adjuvant effect of pain. Although widely used for the treatment of anorexia in palliative care, no randomized clinical trials demonstrating an effect on cancer-associated anorexia, however, in animal models, stimulation of cannabinoid receptors, mainly through CB1 receptor can modulate hypothalamic circuits in the brain stem, which in turn regulate food intake and satiety. Moreover cannabinoids are able to block the effects of TNF in the nervous system, which is associated with appetite changes in cancer patients. Additionally, agonists of cannabinoid receptors attenuated weight loss in murine models of anorexia.

Additionally, to diagnosis anorexia The Anorexia-Cachexia scale (A/CS-12) from The Functional Assessment of Anorexia-Cachexia therapy (FAACT) questionnaire relates differences in symptoms and severity, assigning a value of 0-4 for each of 12 items. A 2010 consensus of special interest group of CACS from ESPEN (The European Society for Clinical Nutrition and Metabolism) in order to unify criteria, proposed that a score ≤24 of the A/CS-12 would be enough to establish a diagnosis of anorexia.

The administration of Nabilone in patients with anorexia associated with Non-Small Cell Lung Cancer (NSCLC) is expected to increase appetite, nutritional status and quality of life.

Methods: randomized double-blind clinical trial assessing Nabilone effect in non-small cell lung cancer (NSCLC) patients with unresectable stage III/IV NSCLC, ECOG performance status (ECOG PS) 1-2 and anorexia (main criteria: score of Anorexia Cachexia scale (AC/S-12) from Functional Assessment of Anorexia Cachexia Therapy ≤24). Patients are randomized to Nabilone at 0.5mg to 1mg, or placebo, given daily orally for 8 weeks. Changes are evaluated from baseline to week 2, 4, and 8.

Time Assessment Dose T0 Baseline 0.5mg T1 2 weeks 1 mg T2 4 weeks 1 mg T3 8 weeks 1 mg

Sample size:

To determine the sample size is considered the effect of cannabinoid (dronabinol, 2.5 mg / 22 days) in appetite in cancer patients by a difference in proportions of 34% more than placebo, requiring 32 patients per group plus 20% of loss gives us a total of 39 patients per group, with a power of 90% and an α of 0.05

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer (NSCLC) patients with unresectable stage IIIB/IV
* ECOG performance status ≤2
* Life expectancy of > 4 months at time of screening
* If woman of childbearing potential or a fertile man, he/she must agree to use an effective form of contraception during the study and for 30 days following the last dose of study drug (an effective form of contraception is abstinence, a hormonal contraceptive, or a double-barrier method)
* Must be willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the protocol tests and procedures

Exclusion Criteria:

* Known allergy to some derivative of marijuana, there is a dependency or who have previously been treated with cannabinoids.
* Consumption of dietary supplements at baseline.
* Currently taking prescription medications intended to increase appetite or treat weight loss; these include, but are not limited to, testosterone, androgenic compounds, megestrol acetate, methylphenidate, and Anamorelin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
anorexia | from the start of consumption until 8 weeks.
  Lack of desire to eat food. Will be obtained through a questionnaire Anorexia / Cachexia scale from Functional Assessment of Anorexia Cachexia Therapy (FAACT) (score ≤24 diagnosis of anorexia)
percentage weight loss | from the start of consumption until 8 weeks.
  percentage weight loss in the last month
Body Mass Index | from the start of consumption until 8 weeks.
  It is an index of a person's weight in relation to height
Subjective Global Assessment | from the start of consumption until 8 weeks.
  convenient, fast and cheaper method used to make a nutritional assessment, consisting of 3 parts: anamnesis, physical examination and qualification.
energy consumption | from the start of consumption until 8 weeks.
  Total calories consumed on average per day for a subject

SECONDARY OUTCOMES:
protein consumption | from the start of consumption until 8 weeks.
  Total protein grams consumed on average per day for a subject
lipids consumption | from the start of consumption until 8 weeks.
  Total lipids grams consumed on average per day for a subject
carbohydrate consumption | from the start of consumption until 8 weeks.
  Total carbohydrate grams consumed on average per day for a subject
nausea | from the start of consumption until 8 weeks.
  adverse effect from Common terminology criteria for adverse event
vomiting | from the start of consumption until 8 weeks.
  adverse effect from Common terminology criteria for adverse event
constipation | from the start of consumption until 8 weeks.
  adverse effect from Common terminology criteria for adverse event
Diarrhea | from the start of consumption until 8 weeks.
  adverse effect from Common terminology criteria for adverse event
Dysgeusia | from the start of consumption until 8 weeks.
  adverse effect from Common terminology criteria for adverse event
Global Status of Quality of Life | from the start of consumption until 8 weeks.
  The Global status of Quality of Life evaluation is evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer with the items 29 and 30.
Physical functioning | from the start of consumption until 8 weeks.
  The Physical functioning evaluation is evaluated from the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer
Role Functioning | from the start of consumption until 8 weeks.
  The Role functioning evaluation is evaluated from the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer
Emotional Functioning | from the start of consumption until 8 weeks.
  The Emotional Functioning evaluation is evaluated from the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer
Social Functioning | from the start of consumption until 8 weeks.
  The Social Functioning evaluation is evaluated from the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer
Nausea/Vomiting | from the start of consumption until 8 weeks.
  The Nausea/Vomiting evaluation is evaluated from the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer
Fatigue | from the start of consumption until 8 weeks.
  The Fatigue evaluation is evaluated from the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer
appetite loss | from the start of consumption until 8 weeks.
  The appetite loss evaluation is evaluated from the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD M Sc, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
publishing the results

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Samet JM. Environmental causes of lung cancer: what do we know in 2003? Chest. 2004 May;125(5 Suppl):80S-3S. doi: 10.1378/chest.125.5_suppl.80s. PMID 15136426
- [Background] Arrieta O, Campos-Parra AD, Zuloaga C, Aviles A, Sanchez-Reyes R, Manriquez ME, Covian-Molina E, Martinez-Barrera L, Meneses A, Cardona A, Borbolla-Escoboza JR. Clinical and pathological characteristics, outcome and mutational profiles regarding non-small-cell lung cancer related to wood-smoke exposure. J Thorac Oncol. 2012 Aug;7(8):1228-34. doi: 10.1097/JTO.0b013e3182582a93. PMID 22659961
- [Background] Watanabe H, Yamamoto N, Tamura T, Shimoyama T, Hotta K, Inoue A, Sawada M, Akiyama Y, Kusaba H, Nokihara H, Sekine I, Kunitoh H, Ohe Y, Kodama T, Saijo N. Study of paclitaxel and dose escalation of cisplatin in patients with advanced non-small cell lung cancer. Jpn J Clin Oncol. 2003 Dec;33(12):626-30. doi: 10.1093/jjco/hyg116. PMID 14769840
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Sarhill N, Mahmoud FA, Christie R, Tahir A. Assessment of nutritional status and fluid deficits in advanced cancer. Am J Hosp Palliat Care. 2003 Nov-Dec;20(6):465-73. doi: 10.1177/104990910302000610. PMID 14649565
- [Background] Arrieta O, Michel Ortega RM, Villanueva-Rodriguez G, Serna-Thome MG, Flores-Estrada D, Diaz-Romero C, Rodriguez CM, Martinez L, Sanchez-Lara K. Association of nutritional status and serum albumin levels with development of toxicity in patients with advanced non-small cell lung cancer treated with paclitaxel-cisplatin chemotherapy: a prospective study. BMC Cancer. 2010 Feb 21;10:50. doi: 10.1186/1471-2407-10-50. PMID 20170547
- [Background] Sanchez-Lara K, Turcott JG, Juarez E, Guevara P, Nunez-Valencia C, Onate-Ocana LF, Flores D, Arrieta O. Association of nutrition parameters including bioelectrical impedance and systemic inflammatory response with quality of life and prognosis in patients with advanced non-small-cell lung cancer: a prospective study. Nutr Cancer. 2012;64(4):526-34. doi: 10.1080/01635581.2012.668744. Epub 2012 Apr 10. PMID 22489794
- [Background] Bossola M, Pacelli F, Doglietto GB. Novel treatments for cancer cachexia. Expert Opin Investig Drugs. 2007 Aug;16(8):1241-53. doi: 10.1517/13543784.16.8.1241. PMID 17685872
- [Background] Wie GA, Cho YA, Kim SY, Kim SM, Bae JM, Joung H. Prevalence and risk factors of malnutrition among cancer patients according to tumor location and stage in the National Cancer Center in Korea. Nutrition. 2010 Mar;26(3):263-8. doi: 10.1016/j.nut.2009.04.013. Epub 2009 Aug 8. PMID 19665873
- [Background] Ross PJ, Ashley S, Norton A, Priest K, Waters JS, Eisen T, Smith IE, O'Brien ME. Do patients with weight loss have a worse outcome when undergoing chemotherapy for lung cancers? Br J Cancer. 2004 May 17;90(10):1905-11. doi: 10.1038/sj.bjc.6601781. PMID 15138470
- [Background] Slaviero KA, Read JA, Clarke SJ, Rivory LP. Baseline nutritional assessment in advanced cancer patients receiving palliative chemotherapy. Nutr Cancer. 2003;46(2):148-57. doi: 10.1207/S15327914NC4602_07. PMID 14690790
- [Background] Muscaritoli M, Anker SD, Argiles J, Aversa Z, Bauer JM, Biolo G, Boirie Y, Bosaeus I, Cederholm T, Costelli P, Fearon KC, Laviano A, Maggio M, Rossi Fanelli F, Schneider SM, Schols A, Sieber CC. Consensus definition of sarcopenia, cachexia and pre-cachexia: joint document elaborated by Special Interest Groups (SIG) "cachexia-anorexia in chronic wasting diseases" and "nutrition in geriatrics". Clin Nutr. 2010 Apr;29(2):154-9. doi: 10.1016/j.clnu.2009.12.004. Epub 2010 Jan 8. PMID 20060626
- [Background] Marin Caro MM, Laviano A, Pichard C. Impact of nutrition on quality of life during cancer. Curr Opin Clin Nutr Metab Care. 2007 Jul;10(4):480-7. doi: 10.1097/MCO.0b013e3281e2c983. PMID 17563467
- [Background] Kosacka M, Werynska B, Golecki M, Jankowska R, Passowicz-Muszynska E. [The incidence and pathogenesis of cancer anorexia-cachexia syndrome in lung cancer]. Pneumonol Alergol Pol. 2008;76(5):360-5. Polish. PMID 19003767
- [Background] Fortunati N, Manti R, Birocco N, Pugliese M, Brignardello E, Ciuffreda L, Catalano MG, Aragno M, Boccuzzi G. Pro-inflammatory cytokines and oxidative stress/antioxidant parameters characterize the bio-humoral profile of early cachexia in lung cancer patients. Oncol Rep. 2007 Dec;18(6):1521-7. PMID 17982639
- [Background] Jatoi A, Qi Y, Kendall G, Jiang R, McNallan S, Cunningham J, Mandrekar S, Yang P. The cancer anorexia/weight loss syndrome: exploring associations with single nucleotide polymorphisms (SNPs) of inflammatory cytokines in patients with non-small cell lung cancer. Support Care Cancer. 2010 Oct;18(10):1299-304. doi: 10.1007/s00520-009-0748-6. Epub 2009 Dec 15. PMID 20012999
- [Background] Laviano A, Meguid MM, Inui A, Muscaritoli M, Rossi-Fanelli F. Therapy insight: Cancer anorexia-cachexia syndrome--when all you can eat is yourself. Nat Clin Pract Oncol. 2005 Mar;2(3):158-65. doi: 10.1038/ncponc0112. PMID 16264909
- [Background] Dewys WD, Begg C, Lavin PT, Band PR, Bennett JM, Bertino JR, Cohen MH, Douglass HO Jr, Engstrom PF, Ezdinli EZ, Horton J, Johnson GJ, Moertel CG, Oken MM, Perlia C, Rosenbaum C, Silverstein MN, Skeel RT, Sponzo RW, Tormey DC. Prognostic effect of weight loss prior to chemotherapy in cancer patients. Eastern Cooperative Oncology Group. Am J Med. 1980 Oct;69(4):491-7. doi: 10.1016/s0149-2918(05)80001-3. PMID 7424938
- [Background] Laviano A, Koverech A, Mari A. Cachexia: clinical features when inflammation drives malnutrition. Proc Nutr Soc. 2015 Nov;74(4):348-54. doi: 10.1017/S0029665115000117. Epub 2015 Mar 26. PMID 25809872
- [Background] Argiles JM, Busquets S, Lopez-Soriano FJ. The pivotal role of cytokines in muscle wasting during cancer. Int J Biochem Cell Biol. 2005 Oct;37(10):2036-46. doi: 10.1016/j.biocel.2005.03.014. PMID 16105746
- [Background] Deans C, Wigmore SJ. Systemic inflammation, cachexia and prognosis in patients with cancer. Curr Opin Clin Nutr Metab Care. 2005 May;8(3):265-9. doi: 10.1097/01.mco.0000165004.93707.88. PMID 15809528
- [Background] LeBlanc TW, Samsa GP, Wolf SP, Locke SC, Cella DF, Abernethy AP. Validation and real-world assessment of the Functional Assessment of Anorexia-Cachexia Therapy (FAACT) scale in patients with advanced non-small cell lung cancer and the cancer anorexia-cachexia syndrome (CACS). Support Care Cancer. 2015 Aug;23(8):2341-7. doi: 10.1007/s00520-015-2606-z. Epub 2015 Jan 14. PMID 25586527
- [Background] Gupta D, Lammersfeld CA, Vashi PG, King J, Dahlk SL, Grutsch JF, Lis CG. Bioelectrical impedance phase angle in clinical practice: implications for prognosis in stage IIIB and IV non-small cell lung cancer. BMC Cancer. 2009 Jan 28;9:37. doi: 10.1186/1471-2407-9-37. PMID 19175932
- [Background] Kubrak C, Jensen L. Critical evaluation of nutrition screening tools recommended for oncology patients. Cancer Nurs. 2007 Sep-Oct;30(5):E1-6. doi: 10.1097/01.NCC.0000290818.45066.00. PMID 17876173
- [Background] Hernandez-Avila M, Romieu I, Parra S, Hernandez-Avila J, Madrigal H, Willett W. Validity and reproducibility of a food frequency questionnaire to assess dietary intake of women living in Mexico City. Salud Publica Mex. 1998 Mar-Apr;40(2):133-40. doi: 10.1590/s0036-36341998000200005. PMID 9617194
- [Background] Thoresen L, Fjeldstad I, Krogstad K, Kaasa S, Falkmer UG. Nutritional status of patients with advanced cancer: the value of using the subjective global assessment of nutritional status as a screening tool. Palliat Med. 2002 Jan;16(1):33-42. doi: 10.1191/0269216302pm486oa. PMID 11963449
- [Background] Berry EM, Mechoulam R. Tetrahydrocannabinol and endocannabinoids in feeding and appetite. Pharmacol Ther. 2002 Aug;95(2):185-90. doi: 10.1016/s0163-7258(02)00257-7. PMID 12182965
- [Background] Touw M. The religious and medicinal uses of Cannabis in China, India and Tibet. J Psychoactive Drugs. 1981 Jan-Mar;13(1):23-34. doi: 10.1080/02791072.1981.10471447. No abstract available. PMID 7024492
- [Background] Davis MP. Oral nabilone capsules in the treatment of chemotherapy-induced nausea and vomiting and pain. Expert Opin Investig Drugs. 2008 Jan;17(1):85-95. doi: 10.1517/13543784.17.1.85. PMID 18095921
- [Background] Osei-Hyiaman D. Endocannabinoid system in cancer cachexia. Curr Opin Clin Nutr Metab Care. 2007 Jul;10(4):443-8. doi: 10.1097/MCO.0b013e3281900ecc. PMID 17563462
- [Background] Pisanti S, Malfitano AM, Grimaldi C, Santoro A, Gazzerro P, Laezza C, Bifulco M. Use of cannabinoid receptor agonists in cancer therapy as palliative and curative agents. Best Pract Res Clin Endocrinol Metab. 2009 Feb;23(1):117-31. doi: 10.1016/j.beem.2009.02.001. PMID 19285265
- [Background] Di Marzo V, Goparaju SK, Wang L, Liu J, Batkai S, Jarai Z, Fezza F, Miura GI, Palmiter RD, Sugiura T, Kunos G. Leptin-regulated endocannabinoids are involved in maintaining food intake. Nature. 2001 Apr 12;410(6830):822-5. doi: 10.1038/35071088. PMID 11298451
- [Background] Walsh D, Nelson KA, Mahmoud FA. Established and potential therapeutic applications of cannabinoids in oncology. Support Care Cancer. 2003 Mar;11(3):137-43. doi: 10.1007/s00520-002-0387-7. Epub 2002 Aug 21. PMID 12618922
- [Background] Kramer JL. Medical marijuana for cancer. CA Cancer J Clin. 2015 Mar;65(2):109-22. doi: 10.3322/caac.21260. Epub 2014 Dec 10. PMID 25503438
- [Result] Cannabis-In-Cachexia-Study-Group; Strasser F, Luftner D, Possinger K, Ernst G, Ruhstaller T, Meissner W, Ko YD, Schnelle M, Reif M, Cerny T. Comparison of orally administered cannabis extract and delta-9-tetrahydrocannabinol in treating patients with cancer-related anorexia-cachexia syndrome: a multicenter, phase III, randomized, double-blind, placebo-controlled clinical trial from the Cannabis-In-Cachexia-Study-Group. J Clin Oncol. 2006 Jul 20;24(21):3394-400. doi: 10.1200/JCO.2005.05.1847. PMID 16849753
- [Result] Foltin RW, Brady JV, Fischman MW. Behavioral analysis of marijuana effects on food intake in humans. Pharmacol Biochem Behav. 1986 Sep;25(3):577-82. doi: 10.1016/0091-3057(86)90144-9. PMID 3774823
- [Result] Plasse TF, Gorter RW, Krasnow SH, Lane M, Shepard KV, Wadleigh RG. Recent clinical experience with dronabinol. Pharmacol Biochem Behav. 1991 Nov;40(3):695-700. doi: 10.1016/0091-3057(91)90385-f. PMID 1666930
- [Result] Nelson K, Walsh D, Deeter P, Sheehan F. A phase II study of delta-9-tetrahydrocannabinol for appetite stimulation in cancer-associated anorexia. J Palliat Care. 1994 Spring;10(1):14-8. PMID 8035251
- [Result] Hart CL, Ward AS, Haney M, Comer SD, Foltin RW, Fischman MW. Comparison of smoked marijuana and oral Delta(9)-tetrahydrocannabinol in humans. Psychopharmacology (Berl). 2002 Dec;164(4):407-15. doi: 10.1007/s00213-002-1231-y. Epub 2002 Sep 14. PMID 12457271
- [Result] Jatoi A, Windschitl HE, Loprinzi CL, Sloan JA, Dakhil SR, Mailliard JA, Pundaleeka S, Kardinal CG, Fitch TR, Krook JE, Novotny PJ, Christensen B. Dronabinol versus megestrol acetate versus combination therapy for cancer-associated anorexia: a North Central Cancer Treatment Group study. J Clin Oncol. 2002 Jan 15;20(2):567-73. doi: 10.1200/JCO.2002.20.2.567. PMID 11786587
- [Result] Woolridge E, Barton S, Samuel J, Osorio J, Dougherty A, Holdcroft A. Cannabis use in HIV for pain and other medical symptoms. J Pain Symptom Manage. 2005 Apr;29(4):358-67. doi: 10.1016/j.jpainsymman.2004.07.011. PMID 15857739
- [Result] Haney M, Rabkin J, Gunderson E, Foltin RW. Dronabinol and marijuana in HIV(+) marijuana smokers: acute effects on caloric intake and mood. Psychopharmacology (Berl). 2005 Aug;181(1):170-8. doi: 10.1007/s00213-005-2242-2. Epub 2005 Oct 15. PMID 15778874
- [Result] Walsh D, Kirkova J, Davis MP. The efficacy and tolerability of long-term use of dronabinol in cancer-related anorexia: a case series. J Pain Symptom Manage. 2005 Dec;30(6):493-5. doi: 10.1016/j.jpainsymman.2005.11.007. No abstract available. PMID 16376734
- [Result] Zutt M, Hanssle H, Emmert S, Neumann C, Kretschmer L. [Dronabinol for supportive therapy in patients with malignant melanoma and liver metastases]. Hautarzt. 2006 May;57(5):423-7. doi: 10.1007/s00105-005-1063-x. German. PMID 16408219
- [Result] Haney M, Gunderson EW, Rabkin J, Hart CL, Vosburg SK, Comer SD, Foltin RW. Dronabinol and marijuana in HIV-positive marijuana smokers. Caloric intake, mood, and sleep. J Acquir Immune Defic Syndr. 2007 Aug 15;45(5):545-54. doi: 10.1097/QAI.0b013e31811ed205. PMID 17589370
- [Result] Maida V, Ennis M, Irani S, Corbo M, Dolzhykov M. Adjunctive nabilone in cancer pain and symptom management: a prospective observational study using propensity scoring. J Support Oncol. 2008 Mar;6(3):119-24. PMID 18402303
- [Result] Brisbois TD, de Kock IH, Watanabe SM, Mirhosseini M, Lamoureux DC, Chasen M, MacDonald N, Baracos VE, Wismer WV. Delta-9-tetrahydrocannabinol may palliate altered chemosensory perception in cancer patients: results of a randomized, double-blind, placebo-controlled pilot trial. Ann Oncol. 2011 Sep;22(9):2086-2093. doi: 10.1093/annonc/mdq727. Epub 2011 Feb 22. PMID 21343383
- [Result] Rowland KM Jr, Loprinzi CL, Shaw EG, Maksymiuk AW, Kuross SA, Jung SH, Kugler JW, Tschetter LK, Ghosh C, Schaefer PL, Owen D, Washburn JH Jr, Webb TA, Mailliard JA, Jett JR. Randomized double-blind placebo-controlled trial of cisplatin and etoposide plus megestrol acetate/placebo in extensive-stage small-cell lung cancer: a North Central Cancer Treatment Group study. J Clin Oncol. 1996 Jan;14(1):135-41. doi: 10.1200/JCO.1996.14.1.135. PMID 8558188
- [Derived] Turcott JG, Del Rocio Guillen Nunez M, Flores-Estrada D, Onate-Ocana LF, Zatarain-Barron ZL, Barron F, Arrieta O. The effect of nabilone on appetite, nutritional status, and quality of life in lung cancer patients: a randomized, double-blind clinical trial. Support Care Cancer. 2018 Sep;26(9):3029-3038. doi: 10.1007/s00520-018-4154-9. Epub 2018 Mar 17. PMID 29550881